CLINICAL TRIAL: NCT06509217
Title: Effects of 12-week Moderate-intensity vs High-intensity Water-aerobic Training on Physical Fitness, Cardiovascular Health, and Well-being in Adults and Older Adults
Brief Title: 12 Weeks of Water Aerobics at Various Intensities for Adults and Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luís Oliveira Brandão Faíl (Other)
Responsible Party: Sponsor-Investigator, Luís Oliveira Brandão Faíl, Guest Assistant, University of Beira Interior
Organization: University of Beira Interior (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ID1475
Record Dates: First submitted 2024-07-11; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Healthy
Keywords: Aquatic exercise; Intensity; Physical fitness; Health-related; Quality of life

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate-intensity Group (Experimental): Participants performed water aerobics at moderate intensities. Water aerobics classes lasted approximately 45 minutes and were held twice a week for 12 weeks
  Interventions: Behavioral: Moderate-intensity Group
- High-intensity Group (Experimental): Participants performed water aerobics at high intensities. Water aerobics classes lasted approximately 45 minutes and were held twice a week for 12 weeks
  Interventions: Behavioral: High-intensity Group

INTERVENTIONS:
Behavioral: Moderate-intensity Group — Water aerobics sessions involved exercises performed at a moderate intensity, between 60% and 70% of the participant's maximum heart rate predicted by their age.
  Arms: Moderate-intensity Group
Behavioral: High-intensity Group — Water aerobics sessions involved exercises performed at a high intensity, between 80% and 90% of the participant's maximum heart rate predicted by their age.
  Arms: High-intensity Group

SUMMARY:
The objective of this clinical trial is to understand the best intensity to perform water aerobics with adults and older adults. The main questions it aims to answer are:

* Is water aerobics performed at high intensity better than water aerobics performed at moderate intensity?
* Is performing water aerobics for 12 weeks good for muscle strength, body composition (body weight, fat mass), lipid profile (triglycerides, cholesterol), blood pressure, and quality of life in adults and older adults?

Participants need:

* Perform water aerobics at high or moderate intensity, twice a week, 45 minutes per class, for 12 weeks
* Be evaluated in the week before starting the water aerobics program (week 0) and at the end week of the program (week 12) regarding muscle strength, body composition, lipid profile, blood pressure, and quality of life

It was hypothesized that independently of the level of intensity used, all variables would improve after water aerobics. It was also expected to observe more gains in all parameters in high-intensity water aerobics compared to moderate intensity

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age

Exclusion Criteria:

* taking part in another physical exercise program
* being recently hospitalized
* having severe motor or cognitive problems
* having any medical restrictions on physical exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in explosive strength of lower limbs at 12 weeks | Baseline and week 12
  The explosive strength of the lower limbs was evaluated using the countermovement jump.Three jumps with countermovement were performed, with participants instructed to jump as high as possible, with one minute of rest between repetitions. A higher jump height corresponds to a better score. In this test, the mean value was considered.
Change from Baseline in explosive strength of upper limbs at 12 weeks | Baseline and week 12
  The explosive strength of the upper limbs was evaluated using medicine ball throw. Each participant was encouraged to throw a 3-kilogram medicine ball, as far as possible. The best scores are achieved by throwing the ball as far as possible. In this test, the mean value was considered.
Change from Baseline in endurance strength of lower limbs at 12 weeks | Baseline and week 12
  The endurance strength of the lower limbs was assessed using the chair stand test. The chair stand test entailed the participant sitting in the center of the chair with a straight back and feet shoulder-width apart and in full contact with the floor. The upper limbs were crossed at the wrist level and positioned against the chest. Upon receiving the starting signal, the participant rose to maximum extension and returned to the initial sitting position, striving to complete the maximum number of repetitions within a 30-second time frame.
Change from Baseline in endurance strength of upper limbs at 12 weeks | Baseline and week 12
  The endurance strength of the upper limbs was assessed using the arm curl test. In this test, the participant was seated in a chair with the back straight and fully leaning against the chair, with their feet flat on the floor. A 2 kg dumbbell was held in their dominant hand, and the test commenced with the forearm in a lower position, near the chair, perpendicular to the floor. Upon receiving the start signal, the participant performed a complete flexion of the forearm and then returned to the initial position of forearm extension. The evaluator encouraged the participant to perform as many repetitions as possible within a time limit of 30 seconds, counting each correct flexion performed.
Change from Baseline in body mass at 12 weeks | Baseline and week 12
  A bioimpedance balance was used. For the correct extraction of this test, participants were barefoot and dressed in as little clothing as possible.
Change from Baseline in fat mass percentage at 12 weeks | Baseline and week 12
Change from Baseline in fat-free mass at 12 weeks | Baseline and week 12
Change from Baseline in body mass index at 12 weeks | Baseline and week 12
  The body mass index (BMI) was calculated by dividing the body mass value by the height squared (kg/m^2). For this, each participant's height was measured using a precision stadiometer with a scale of 0.001 m. For the correct extraction of this test, participants were barefoot.
Change from Baseline in triglycerides at 12 weeks | Baseline and week 12
  Blood samples were collected before exercise (after a 15-minute rest period) and at least 2 hours after the last meal.
Change from Baseline in total cholesterol at 12 weeks | Baseline and week 12
Change from Baseline in diastolic blood pressure at 12 weeks | Baseline and week 12
  This measure was assessed using an automatic blood pressure monitor, after the participant was seated and resting for at least 20 minutes.
Change from Baseline in systolic blood pressure at 12 weeks | Baseline and week 12
Change from Baseline in resting heart rate at 12 weeks | Baseline and week 12
  This measure was assessed using an automatic blood pressure monitor, after the participant was seated and resting for at least 20 minutes.

SECONDARY OUTCOMES:
Change from Baseline in quality of life at 12 weeks | Baseline and week 12
  The WHOQOL-BREF (Portuguese version) questionnaire with 26 items was used to assess the participants' quality of life. Of the 26 items, 2 are related to the general quality of life and general health, and the remaining 24 items assess the perception of quality of life in 4 domains: physical, psychological, social relationships, and environment. The higher the final score, the higher the participant's quality of life in each domain.

CONTACTS AND LOCATIONS:
Overall Officials: Luís Faíl, Principal Investigator — University of Beira Interior
Locations (1):
- Tramagal Municipal Swimming Pool, Abrantes, Portugal

IPD SHARING:
Plan to Share IPD: No